CLINICAL TRIAL: NCT02342470
Title: A Multi-center, Randomized, Double-blind, Parallel, Placebo-controlled, Dose-finding, Phase IIa Clinical Trial to Efficacy and Safety of PMK-S005 for the Prevention of Recurrent Peptic Ulcer in Low-dose Aspirin Users
Brief Title: Efficacy and Safety of PMK-S005 in the Prevention of Recurrent Peptic Ulcer in Low-dose Aspirin Users
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PharmaKing (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PMK-S005_Phase II
Record Dates: First submitted 2014-12-19; First posted 2015-01-21 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Peptic Ulcer
Keywords: prevention; Recurrent peptic ulcer
MeSH Terms: conditions — Peptic Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo Comparator / Bid
  Interventions: Drug: Placebo
- PMK-S005 1 (Experimental): Total 50mg, by mouth, bid
  Interventions: Drug: PMK-S005 1
- PMK-S005 2 (Experimental): Total 100mg, by mouth, bid
  Interventions: Drug: PMK-S005 2
- PMK-S005 3 (Experimental): Total 150mg, by mouth, bid
  Interventions: Drug: PMK-S005 3

INTERVENTIONS:
Drug: Placebo — Drug : Placebo
  Arms: Placebo
Drug: PMK-S005 1 — Drug : PMK-S005 1 (50mg)
  Arms: PMK-S005 1
Drug: PMK-S005 2 — Drug : PMK-S005 2 (100mg)
  Arms: PMK-S005 2
Drug: PMK-S005 3 — Drug : PMK-S005 3 (150mg)
  Arms: PMK-S005 3

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety by comparing prevention of recurrent peptic ulcer in low-dose aspirin users between PMK-S005 and Placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 19 years of age
* Accompanied by hypertension, diabetes, ischemic heart disease, arrhythmia, dyslipidemia patients who are required to continuous administration of low-dose aspirin(100mg)
* Patients who get Modified Lanza Score (MLS) 0 in screening period according to endoscopic findings
* Patients who have stomach or duodenal ulcer scar in screening period according to endoscopic findings. But, the cases that scars caused by other disorders or endoscopic treatment are excluded
* Patients who have no digestive symptoms(except for mild physconia, abdominal pain, diarrhea and vomit, nausea-vomiting) in screening period
* Signature of the written informed consent

Exclusion Criteria:

* Within 4 weeks prior to screening period, patients who continuously take aspirin or NSAIDs
* Patient who has hypersensitivity to PMK-S005 and aspirin components or is banned to use them
* Patients who had a abdominal surgery that affect gastrointestinal motility (Except appendectomy and hysterectomy), But, patients who had enterectomy is excluded regardless of the time period
* Patients who are judged by investigator that they have other upper gastroesophageal disease, active/healing-stage peptic ulcer, digestive malignant tumor or Barrett's esophagus
* Patients with Irritable Bowel Syndrome (IBS), Inflammatory Bowel Disease (IBD), Ulcerative Colitis, Crohn's disease, Zolinger-Ellison syndrome
* History of esophagus, liver, pancreas, stomach, colorectal cancer or malignant tumors within 5 years
* History of malabsorption within 3 months prior to screening period
* Patients who have been taken drug that affect the validity within 2 weeks before beginning of the clinical test
* Patient who is needed continuously to take antithrombotic agents , anti- coagulant , anti- choline agents, prostaglandins , mucosal protective agents , methotrexate, antidepressants , iron treat agents during clinical test.
* Patients with clinical meaningful laboratory test results
* Known alcohol and/or any other drug abuse or dependence
* Pregnant or lactating women
* Women planning to become pregnant
* Within 1 month, patients who have been taken other clinical test drug
* Patients who are judged by investigator that participation of the study is difficult

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2014-11-24 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2017-12-08 (Actual)

PRIMARY OUTCOMES:
The incidence of endoscopic peptic ulcer | 12 weeks

SECONDARY OUTCOMES:
The incidence of endoscopic stomach / duodenal mucosal disease(erosion, ulcer) | 12 weeks
The incidence of endoscopic stomach / duodenal erosion | 12 weeks
The incidence of endoscopic stomach / duodenal ulcer | 12 weeks
The changes of MLS in the gastroduodenal endoscopy result compared to baseline | 12 weeks
The incidence of endoscopic esophagitis | 16 weeks
Rescue drug use count and the total amount | 16 weeks
Changes in gastrointestinal symptoms score | 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Bundang Seoul University Hospital, Kumi-dong, Bundang-gu, Seongnam-si, Gyeonggi-do, South Korea